CLINICAL TRIAL: NCT04605198
Title: Mindfulness-based Intervention to Address PTSD in Trauma-exposed, Homeless Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Dana Rose Garfin, Assistant Adjunct Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-5607; 5K01MD013910 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Stress Disorders, Post-Traumatic; Depressive Symptoms; Hydrocortisone; Substance Use
Keywords: PTSD; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Substance-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from two sites. To avoid contamination between subjects living at the sites, using a quasi-randomized method, all participants at each site will receive the same treatment per cohort. Sites will alternate between the assignment of treatment (modified-MBSR) or control (health promotion class) in sequential cohorts to account for between site differences.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Mindfulness-based Stress Reduction (Experimental)
  Interventions: Behavioral: Modified Mindfulness-based Stress Reduction
- Health Promotion Attention Control (Active Comparator)
  Interventions: Behavioral: Health Promotion Wellness Classes

INTERVENTIONS:
Behavioral: Modified Mindfulness-based Stress Reduction — Participants will be trained in mindfulness meditation and the applicability of mindfulness practices to daily life. During MBSR programming, teachers will lecture about key topics in mindfulness and lead class discussions. Participants are given homework assignments, such as listening to guided meditations. Participants are given opportunities to ask the instructor questions and to share their experiences with each other. Each session focuses on a different key topic. Topics are: Session 1: Introduction; Session 2: Understanding Perceptions; Session 3: Hatha Yoga, Sitting Meditation, Walking Meditation; Session 4: Concentration & Awareness; Session 5: Unhealthy Patterns &Getting Unstuck; Session 6: Transformational Coping Strategies; Session 7: Mini-retreat; Session 8: Maintaining Discipline & Flexibility; Session 9: Course Review.
  Other Names: modified MBSR
  Arms: Modified Mindfulness-based Stress Reduction
Behavioral: Health Promotion Wellness Classes — Sessions will cover the following general wellness topics: Session 1; Introduction; Session 2: Envisioning Health Through Art; Session 3: Chronic Disease 1 (Heart Health); Session 4: Chronic Disease II (Diabetes); Session 5: Nutrition and Hydration; Session 6: Infectious Disease Prevention; Session 7: Skin Care; Session 8: Oral Health; Session 9: Promoting Social Integration & Course Graduation.
  Arms: Health Promotion Attention Control

SUMMARY:
Posttraumatic stress disorder (PTSD) is a major public health concern that disproportionately effects minorities and those with low-socioeconomic status, such as homeless women, creating a critical health disparity. PTSD has been linked with dysregulated hypothalamic-pituitary-adrenal (HPA) functioning and increased inflammation, which can lead to long-term physical-health problems and PTSD-symptom maintenance, exacerbating disparities. Mindfulness-based interventions, including Mindfulness-based Stress Reduction (MBSR), have shown promise as a complementary tool for addressing PTSD in veterans and with low-income, minority populations, but homeless women have not been examined adequately. MBSR may improve PTSD symptomatology and help modulate the dysregulated stress response common in individuals with PTSD, improving physical and mental health concurrently. This project is an open-label, parallel, modified-cross over clinical trial of a modified-MBSR intervention to reduce PTSD symptoms in homeless women and to explore physiological correlates of treatment-response.

Hypotheses:

1. Participation in an MBSR-based intervention will be associated with clinically significant reduction in PTSD (primary outcome), lower depression symptoms and greater drug and alcohol abstinence (secondary outcomes) compared to participation in an attention control.
2. Compared to an attention control, participants in an MBSR-based intervention group will demonstrate improvements in cortisol reactivity and lower inflammation.

At baseline, women will complete psychosocial assessments (e.g., depression, substance use, trauma history) and participate in a brief stress task, providing salivary samples before and after the task (which will be assayed for cortisol and C-reactive protein, a marker of inflammation). Women will then participate in 1) a 9-session MBSR-based program that was modified based on an initial qualitative component that involved a Community Advisory Board and focus groups with women from the community (N=4 focus groups; 28 women total) or 2) a nine-session health-promotion course (i.e., attention-control condition). Follow-up assessments that include psychosocial and biological data will occur immediately after final intervention session and again 6-months later. Clinically-meaningful improvements in PTSD (primary outcome) and secondary outcomes (e.g., depression, substance use, inflammation, cortisol reactivity) will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. self-reported homeless women
2. age 18+
3. willing to provide informed consent
4. lifetime exposure to at least one Diagnostic and Statistical Manuel of Mental Disorders, version 5 (DSM-5) qualifying trauma
5. likely subthreshold or threshold PTSD, as measured by the PTSD Checklist for Civilians for DSM-5.

Note: A homeless person is defined as anyone who spent the previous night in a public or private shelter, or on the street.

Exclusion Criteria:

1. not speaking English
2. judged to be cognitively impaired; as indicated by score >9 on the Short-Blessed Screener (SBS).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women are eligible for the study.
Enrollment: 156 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - North County Serenity House, Escondido, California
  - Prototypes Women's Center, Pomona, California

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 192 participants were assessed for eligibility. Of those, 13 did not experience homelessness, 10 were cognitively impaired, 3 did not meet criteria for subthreshold PTSD, and 10 were eligible but did not enroll.
Groups:
- Modified Mindfulness-based Stress Reduction (MBSR): Modified Mindfulness-based Stress Reduction (MBSR): Participants will be trained in mindfulness meditation and the applicability of mindfulness practices to daily life. During MBSR programming, teachers will lecture about key topics in mindfulness and lead class discussions. Participants are given homework assignments, such as listening to guided meditations. Participants are given opportunities to ask the instructor questions and to share their experiences with each other. Each session focuses on a different key topic. Topics are: Session 1: Introduction; Session 2: Understanding Perceptions; Session 3: Hatha Yoga, Sitting Meditation, Walking Meditation; Session 4: Concentration & Awareness; Session 5: Unhealthy Patterns &Getting Unstuck; Session 6: Transformational Coping Strategies; Session 7: Mini-retreat; Session 8: Maintaining Discipline & Flexibility; Session 9: Course Review.
- Health Promotion Attention Control (HP Control): Health Promotion Wellness Classes: Sessions will cover the following general wellness topics: Session 1; Introduction; Session 2: Envisioning Health Through Art; Session 3: Chronic Disease 1 (Heart Health); Session 4: Chronic Disease II (Diabetes); Session 5: Nutrition and Hydration; Session 6: Infectious Disease Prevention; Session 7: Skin Care; Session 8: Oral Health; Session 9: Promoting Social Integration & Course Graduation.
Period: Overall Study
Arm/Group | Modified Mindfulness-based Stress Reduction (MBSR) | Health Promotion Attention Control (HP Control)
Started | 90 | 66
Completed | 71 | 47
Not Completed | 19 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Mindfulness-based Stress Reduction | Health Promotion Attention Control | Total
Number analyzed (Participants) | 90 | 66 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.52 (9.79) | 35.18 (11.23) | 35.38 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 66 | 156
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 29 | 79
  Not Hispanic or Latino | 40 | 37 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 16 | 33
  Black/African American | 20 | 13 | 33
  Hispanic | 43 | 23 | 66
  Mixed identity | 2 | 4 | 6
  Native American/Pacific Islander | 8 | 10 | 18
Posttraumatic Stress Disorder Checklist for Diagnostic & Statistical Manual of Mental Disorders, 5th [Mean (Standard Deviation); unit: units on a scale] — The Posttraumatic Stress Disorders Checklist for Diagnostic and Statistical Manuel of Mental Disorders, 5th Edition (PCL-5) first identifies prior direct exposure to a DSM-V traumatic event. Then, twenty items assess all four B-E criteria (re-experiencing, avoidance, negative thoughts or cognitions, hyperarousal), on scale from 0=not at all to 4=extremely. The range of symptoms is 0-80. Thirty-three is generally considered the cutpoint for probable-PTSD.
  units on a scale | 40.40 (16.44) | 47.46 (14.63) | 45.70 (15.72)
Mean PROMIS Depression [Mean (Standard Deviation); unit: units on a scale] — The Patient-Reported Outcomes Measurement Information System (PROMIS), Depression, Short Form assesses frequency of eight symptoms of depression in the past seven days from 1=never to 5=always. The range is 8-40.
  units on a scale | 17.72 (8.28) | 20.42 (8.80) | 18.87 (8.58)
Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety [Mean (Standard Deviation); unit: units on a scale] — The Patient-Reported Outcomes Measurement Information System (PROMIS), Anxiety Short Form assesses frequency of seven symptoms of anxiety in the past seven days from 1=never to 5=always. The range is 7-35.
  units on a scale | 20.88 (6.67) | 22.12 (7.04) | 21.40 (6.84)
Substance Use - Texas Christian University Drug Screen [Mean (Standard Deviation); unit: units on a scale] — The Texas Christian University Drug Screen (TCU Drug Screen 5) is a 19-item screener for Diagnostic and Statistical Manual of Mental Disorders criteria substance use disorder. For the first 13 items, participants indicate 0=no or 1=yes. To score, assign 1 point to each "yes" response to items 1 through 9. For items 10 and 11, a. assign 1 point if respondent answers "yes" to either 10a or 10b; b. assign 1 point if respondent answers "yes" to either 11a or 11b. 3. Sum 1-point "yes" responses for items 1 to11, yielding a total score range 0 to 11. The remaining items are not scored.
  units on a scale | 8.68 (2.40) | 8.98 (2.45) | 8.81 (2.42)
Substance use, 5-panel test [Count of Participants; unit: Participants] — 5-panel substance use urine test (tests for amphetamine, cocaine, methamphetamine, opioids, and THC), coded 0=no drugs in urine, 1=at least one substance in urine
  Participants | 9 | 2 | 11
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)] | 4639.62 (9332.93) | 1330.49 (2160.09) | 3239.60 (7393.32)
Cortisol reactivity [Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)] — At baseline, participants engaged in a stress task (trauma script imagery test). Participants provided cortisol samples via passive saliva drool before and then twenty minutes post-task. Baseline cortisol reactivity was calculated by subtracting pre-task cortisol from the post-task cortisol. To collect saliva, participants passively drooled into a collection vial for three minutes or until 0.80 milliliters of fluid was collected. Saliva samples were immediately placed in the on-site freezer and subsequently frozen at -80°C until assayed Population: Some data was contaminated or did not have adequate volume for analyses, thus 144 rather than 156 observations were available.
  Milligrams per deciliter (mg/dL)
    number analyzed (Participants) | 84 | 60 | 144
    (all) | -.912 (2.32) | -.617 (2.41) | -.789 (2.35)

OUTCOME MEASURES:

1. Primary Outcome: Post-traumatic Stress Symptoms (PTSD) as Measured by the PTSD Checklist for DSM 5 (PCL-5) (DSM=Diagnostic and Statistical Manuel of Mental Disorders).
Description: Change in Posttraumatic Stress Symptoms Disorder symptoms (i.e., decrease in symptoms), as measured by the PTSD Checklist for DSM 5 (PCL-5) (DSM=Diagnostic and Statistical Manuel of Mental Disorders). The PCL-5 is a 20-item scale (range 0-80), with rating scale descriptions: 0 "Not at all," 1 "A little bit," 2 "Moderately," 3 "Quite a bit," and 4 "Extremely." Higher scores indicate more PTSD symptoms.
Time Frame: Immediately post-intervention & 6-month follow-up
Population: The total number analyzed for Time 2 (immediate post-intervention follow-up) was 125. The total number analyzed for Time 3 was 86. The numbers differ due to attrition over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Mindfulness-based Stress Reduction | Health Promotion Attention Control
Number analyzed (Participants) | 73 | 52
score on a scale
  Time 2 (immediate post-intervention) | 26.93 (18.20) | 30.75 (16.62)
  Time 3 (6-month follow-up): number analyzed (Participants) | 50 | 36
  Time 3 (6-month follow-up) | 24.46 (15.38) | 28.33 (14.88)
Statistical Analysis 1: Comparison: Modified Mindfulness-based Stress Reduction vs Health Promotion Attention Control; Test type: Superiority — A multilevel model was constructed. Participants were entered as random effects to nest observations within participants. Group assignment (i.e., MBSR vs. Health Promotion Control), time (i.e., Time 1 [baseline], Time 2 [immediate post-intervention, primary endpoint], and Time 3 [6-month follow-up]), and group-by-time interactions were entered as fixed effects. Site was also included as a fixed-effect. An independent covariance pattern was specified as final models were random-intercept only; p = .846, Mixed Models Analysis; Mean Difference (Net) = -0.58, 95% CI 2-sided [-6.46 to 5.29] — The estimate represents the interaction term for group by time interaction for the immediate follow-up, with the control group coded 0 and the intervention group coded as 1

2. Secondary Outcome: Depression
Description: Change in depressive symptoms from baseline to follow-ups (i.e., decrease in symptoms), using the Patient Reported Outcomes Measurement Information System (PROMIS) measure for depression. The PROMIS asks 9-items (range 9-45) with response options: 1 "never", 2 "rarely", 3 "sometimes", 4 "often", and 5 "always". Higher scores indicate more symptoms of depression.
Time Frame: Immediately post-intervention & 6-month follow-up
Population: The total number analyzed for Time 2 (immediate post-intervention follow-up) was 126. The total number analyzed for Time 3 was 86. The numbers differ due to attrition over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Mindfulness-based Stress Reduction | Health Promotion Attention Control
Number analyzed (Participants) | 73 | 53
score on a scale
  Time 2 (immediate post-intervention) | 13.19 (6.52) | 17.98 (8.24)
  Time 3 (6-month follow-up): number analyzed (Participants) | 50 | 36
  Time 3 (6-month follow-up) | 11.98 (5.06) | 16.97 (6.66)
Statistical Analysis 1: Comparison: Health Promotion Attention Control; A multilevel model was constructed. Participants were entered as random effects to nest observations within participants. Group assignment (i.e., MBSR vs. Health Promotion Control), time (i.e., Time 1 [baseline], Time 2 [immediate post-intervention, primary endpoint], and Time 3 [6-month follow-up]), and group-by-time interactions were entered as fixed effects. Site was also included as a fixed-effect. An independent covariance pattern was specified as final models were random-intercept only; Test type: Superiority; p = .139, Mixed Models Analysis; Mean Difference (Net) = -1.88, 95% CI 2-sided [-4.36 to 0.60] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Substance Use Measured by the Texas Christian University Screen for Diagnostic and Statistical Manuel of Mental Disorders, 5th Edition (TCU 5)
Description: Change in continues measure of self-report substance use from baseline to follow-ups using the Texas Christian University Screen for Diagnostic and Statistical Manuel of Mental Disorders, 5th Edition (TCU 5). The possible range for the score is 1-11. Participants respond to a series of 13 possible no (0) or yes (1) questions, with two questions counting for a maximum score of "1" each. Higher scores indicate more severe substance use.
Time Frame: Immediately post-intervention & 6-month follow-up
Population: The total number analyzed for Time 2 (immediate post-intervention follow-up) was 119. The total number analyzed for Time 3 was 86. The numbers differ due to attrition and missing data over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Mindfulness-based Stress Reduction | Health Promotion Attention Control
Number analyzed (Participants) | 90 | 66
score on a scale
  Time 2 (immediate post-intervention): number analyzed (Participants) | 73 | 46
  Time 2 (immediate post-intervention) | 0.68 (1.79) | 1.71 (2.56)
  Time 3 (6-month follow-up): number analyzed (Participants) | 50 | 36
  Time 3 (6-month follow-up) | 1.24 (2.43) | 1.28 (3.05)
Statistical Analysis 1: Comparison: Health Promotion Attention Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .222, Mixed Models Analysis; Mean Difference (Net) = -0.12, 95% CI 2-sided [-1.21 to 0.97] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Positive Substance Use Measured by a 5-panel FDA-approved Urine Test Cup
Description: Count of participants with positive substance use from baseline to follow-up using 5-panel FDA-approved urine test cup.
Time Frame: Immediately post-intervention & 6-month follow-up
Population: The total number analyzed for Time 2 (immediate post-intervention follow-up) was 118. The total number analyzed for Time 3 was 79. The numbers differ due to attrition and missing data over time.
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Mindfulness-based Stress Reduction | Health Promotion Attention Control
Number analyzed (Participants) | 71 | 47
Participants
  Time 2 (immediate post-intervention); total number positive for any substance | 4 | 3
  Time 3 (6-month follow-up); total number positive for any substance: number analyzed (Participants) | 48 | 31
  Time 3 (6-month follow-up); total number positive for any substance | 2 | 3
Statistical Analysis 1: Comparison: Health Promotion Attention Control; A multilevel model was constructed using a logit distribution. Participants were entered as random effects to nest observations within participants. Group assignment (i.e., MBSR vs. Health Promotion Control), time (i.e., Time 1 [baseline], Time 2 [immediate post-intervention], and Time 3 [6-month follow-up]), and group-by-time interactions were entered as fixed effects. Site was included as a fixed-effect. An independent covariance pattern was specified. Final models were random-intercept only; Test type: Superiority; p = 0.166, Mixed Models Analysis; Odds Ratio, log = -1.76, 95% CI 2-sided [-4.26 to 0.73] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Cortisol Reactivity
Description: Change in cortisol reactivity using script driven imagery from baseline to follow-up using standard manufacturer protocols (from Salimetrics). Higher scores indicate more change in cortisol.
Time Frame: Immediately post-intervention & 6-month follow-up
Population: The total number analyzed for Time 2 (immediate post-intervention follow-up) was 118. The total number analyzed for Time 3 was 76. The numbers differ due to attrition and missing data over time.
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (µg/dL)
Arm/Group | Modified Mindfulness-based Stress Reduction | Health Promotion Attention Control
Number analyzed (Participants) | 71 | 47
Micrograms per deciliter (µg/dL)
  Time 2 (immediate post-intervention) | -2.10 (10.45) | -0.70 (3.98)
  Time 3 (6-month follow-up): number analyzed (Participants) | 46 | 30
  Time 3 (6-month follow-up) | -2.45 (10.53) | -1.76 (9.11)
Statistical Analysis 1: Comparison: Health Promotion Attention Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .737, Mixed Models Analysis; Mean Difference (Net) = -0.52, 95% CI 2-sided [-3.57 to 2.53] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: C-Reactive Protein (CRP)
Description: Change in CRP, measured via saliva using the Salivary C-Reactive Protein ELISA kit, an enzyme-linked immunoassay. Higher scores indicate higher concentration of CRP.
Time Frame: Immediately post-intervention & 6-month follow-up
Population: The total number analyzed for Time 2 (immediate post-intervention follow-up) was 121. The total number analyzed for Time 3 was 80. The numbers differ due to attrition and missing data over time.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Modified Mindfulness-based Stress Reduction | Health Promotion Attention Control
Number analyzed (Participants) | 72 | 49
Milligrams per deciliter (mg/dL)
  Time 2 (immediate post-intervention) | 2395.32 (3542.12) | 1725.80 (3266.13)
  Time 3 (6-month follow-up): number analyzed (Participants) | 48 | 32
  Time 3 (6-month follow-up) | 3950.69 (7617.19) | 1248.06 (1390.65)
Statistical Analysis 1: Comparison: Health Promotion Attention Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .024, Mixed Models Analysis; Mean Difference (Net) = -2391.98, 95% CI 2-sided [-4471.46 to -312.49] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the duration of the intervention procedures (approximately 8 weeks).
Arm/Group | Modified Mindfulness-based Stress Reduction | Health Promotion Attention Control
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/66
Other Adverse Events (participants affected / at risk) | 0/90 | 0/66

LIMITATIONS AND CAVEATS:
Participants were not assigned on a 1:1 ratio. Some courses lasted more than 8 weeks due to vacillating quarantines and lockdowns during COVID-19 outbreaks. Relatedly, participants who were discharged from the site were not allowed to participate in follow-up sessions due to COVID-19 quarantines in 2020-2021, contributing to increased attrition over time. Additional MBSR participants were enrolled to adjust for this, allowing for adequate power but resulting in an unbalanced design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04605198/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT04605198/ICF_000.pdf